CLINICAL TRIAL: NCT01283139
Title: A Phase 2b, Dose-ranging Study to Evaluate the Efficacy and Safety of Sifalimumab in Adults With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Efficacy and Safety of Sifalimumab in Adults With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-IA-MEDI-545-1067; 2010-024069-30 (EudraCT Number)
Record Dates: First submitted 2011-01-20; First posted 2011-01-25 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Systemic Lupus Erythematosus; Sifalimumab; MEDI-545
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — sifalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sifalimumab 200 milligram (mg) (Experimental): Sifalimumab 200 milligram (mg) will be administered intravenously every 2 weeks for 4 weeks and then monthly for 44 weeks for a total of 14 doses.
  Interventions: Biological: Sifalimumab 200 mg
- Sifalimumab 600 mg (Experimental): Sifalimumab 600 mg will be administered intravenously every 2 weeks for 4 weeks and then monthly for 44 weeks for a total of 14 doses.
  Interventions: Biological: Sifalimumab 600 mg
- Sifalimumab 1,200 mg (Experimental): Sifalimumab 1,200 mg will be administered intravenously every 2 weeks for 4 weeks and then monthly for 44 weeks for a total of 14 doses.
  Interventions: Biological: Sifalimumab 1,200 mg
- Placebo (Placebo Comparator): Placebo matching to sifalimumab will be administered intravenously at a fixed dose every 2 weeks for 4 weeks and then monthly for 44 weeks for a total of 14 doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sifalimumab 200 mg — Sifalimumab 200 mg intravenously every 2 weeks for 4 weeks and then monthly for 44 weeks for a total of 14 doses.
  Other Names: MEDI-545
  Arms: Sifalimumab 200 milligram (mg)
Biological: Sifalimumab 600 mg — Sifalimumab 600 mg intravenously every 2 weeks for 4 weeks and then monthly for 44 weeks for a total of 14 doses.
  Other Names: MEDI-545
  Arms: Sifalimumab 600 mg
Biological: Sifalimumab 1,200 mg — Sifalimumab 1,200 mg intravenously every 2 weeks for 4 weeks and then monthly for 44 weeks for a total of 14 doses.
  Other Names: MEDI-545
  Arms: Sifalimumab 1,200 mg
Other: Placebo — IV Placebo every 2 weeks for 4 weeks and then monthly for 44 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of sifalimumab compared to placebo in subjects with moderately to severely active Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase 2b, multinational, multicenter, randomized, double-blind, placebo controlled, parallel group study to evaluate the efficacy and safety of three intravenous (IV) treatment regimens of sifalimumab (200, 600, or 1,200 mg) in adult subjects with chronic moderately-to-severely active SLE with an inadequate response to standard of care (SOC) for SLE.

ELIGIBILITY:
Inclusion Criteria: - Fulfills at least 4 of American College of Rheumatology (ACR) criteria for systemic lupus erythematosus (SLE) including a positive antinuclear antibody (ANA) or elevated ds-deoxyribonucleic acid (DNA) or Sm antibody at screening - Disease history of SLE greater than or equal to (>=) 24 weeks at screening - Weight more than (>) 40 kilogram (kg) - Currently receiving stable dose of oral prednisone and/or antimalarials/immunosuppressives - Active moderate to severe SLE disease based on SLE disease activity score (SLEDAI) and British Isles Lupus Assessment Group Index (BILAG) and Physicians Global Assessment - No evidence of cervical malignancy on PAP within 6 months of randomization - Female subjects must be willing to avoid pregnancy - Negative TB test or newly positive TB test due to latent TB for which treatment must be initiated at or before randomization. Exclusion Criteria: - Active severe SLE-driven renal disease or unstable renal disease prior to screening - Active severe or unstable neuropsychiatric SLE - Clinically significant active infection including ongoing and chronic infections - History of human immunodeficiency virus (HIV) - Confirmed Positive tests for Hepatitis B or positive test for hepatitis C - History of severe herpes infection such as herpes encephalitis, ophthalmic herpes, disseminated herpes - Herpes Zoster within 3 months of screening - History of cancer other than basal cancer or cervical cancer treated with apparent success >=1 year prior to randomization - Receipt of a biologic agent within 5 half-lives or prior to loss of pharmacodynamic and/or clinical effect (whichever is longer) prior to screening - Live or attenuated vaccine within 4 weeks prior to screening - Subjects with substance abuse - Subjects with significant hematologic abnormalities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2013-11-14 (Actual); Study Completion 2014-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Illei, MD, Study Director — MedImmune LLC
Locations (107):
- United States (17):
  - Research Site, La Jolla, California
  - Research Site, Palm Desert, California
  - Research Site, San Leandro, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Orlando, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Lansing, Michigan
  - Research Site, Brooklyn, New York
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Dallas, Texas
  - Research Site, Seattle, Washington
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Quilmes
  - Research Site, San Miguel de Tucumán
- Brazil (6):
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Juiz de Fora
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (2):
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Chile (3):
  - Research Site, Osorno
  - Research Site, Santiago
  - Research Site, Viña del Mar
- France (4):
  - Research Site, Bordeaux
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Paris
  - Research Site, Strasbourg
- Germany (10):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Regensburg
  - Research Site, Würzburg
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Zalaegerszeg
- India (2):
  - Research Site, Bangalore
  - Research Site, Secunderabad
- Italy (6):
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Roma
- Research Site, Kingston, Jamaica
- Mexico (4):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, San Luis Potosí City
- Research Site, Amsterdam, Netherlands
- Peru (2):
  - Research Site, Lima
  - Research Site, San Borja
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Iloilo City
  - Research Site, Manila
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Tg Mures
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pinelands
  - Research Site, Soweto
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Guadalajara
  - Research Site, La Laguna (Tenerife)
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- Research Site, Bangkok, Thailand
- United Kingdom (7):
  - Research Site, Brighton
  - Research Site, Cambridge
  - Research Site, Cannock
  - Research Site, Guildford
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Background] Khamashta M, Merrill JT, Werth VP, Furie R, Kalunian K, Illei GG, Drappa J, Wang L, Greth W; CD1067 study investigators. Sifalimumab, an anti-interferon-alpha monoclonal antibody, in moderate to severe systemic lupus erythematosus: a randomised, double-blind, placebo-controlled study. Ann Rheum Dis. 2016 Nov;75(11):1909-1916. doi: 10.1136/annrheumdis-2015-208562. Epub 2016 Mar 23. PMID 27009916
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Brohawn PZ, Streicher K, Higgs BW, Morehouse C, Liu H, Illei G, Ranade K. Type I interferon gene signature test-low and -high patients with systemic lupus erythematosus have distinct gene expression signatures. Lupus. 2019 Nov;28(13):1524-1533. doi: 10.1177/0961203319885447. Epub 2019 Oct 29. PMID 31660791

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 834 participants were screened out of which 402 participants did not meet eligibility criteria and were considered screen failures, and 432 participants were randomized into the study.
Groups:
- Placebo: Placebo matching to sifalimumab administered by intravenous infusion at a fixed dose of every 2 weeks (14 days) for the first 3 doses (Days 1, 15, and 29) and then every 4 weeks (28 days) thereafter for 11 doses for a total of 14 doses.
- Sifalimumab 200 Milligram (mg): Sifalimumab 200 mg administered by intravenous infusion every 2 weeks (14 days) for the first 3 doses (Days 1, 15, and 29) and then every 4 weeks (28 days) thereafter for 11 doses for a total of 14 doses.
- Sifalimumab 600 mg: Sifalimumab 600 mg administered by intravenous infusion every 2 weeks (14 days) for the first 3 doses (Days 1, 15, and 29) and then every 4 weeks (28 days) thereafter for 11 doses for a total of 14 doses.
- Sifalimumab 1,200 mg: Sifalimumab 1,200 mg administered by intravenous infusion every 2 weeks (14 days) for the first 3 doses (Days 1, 15, and 29) and then every 4 weeks (28 days) thereafter for 11 doses for a total of 14 doses.
Period: Overall Study
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Started | 108 | 108 | 109 | 107
Completed | 91 | 90 | 91 | 92
Not Completed | 17 | 18 | 18 | 15
Not completed — Lost to Follow-up | 5 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 8 | 8 | 6 | 8
Not completed — Death | 2 | 0 | 2 | 2
Not completed — Lack of Efficacy | 1 | 2 | 2 | 1
Not completed — Early termination due to AE/SAE | 1 | 1 | 0 | 0
Not completed — Participant's refusal to continue | 0 | 3 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Missed follow-up visit | 0 | 1 | 2 | 2
Not completed — Participant randomized in error | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg | Total
Number analyzed (Participants) | 108 | 108 | 109 | 107 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (12.3) | 39.9 (11.4) | 40.1 (11.3) | 39.4 (12.1) | 39.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 103 | 98 | 97 | 399
  Male | 7 | 5 | 11 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Response in Systemic Lupus Erythematosus Responder Index 4 (SRI [4])
Description: SRI (4) responder is defined as: 1) a reduction in baseline Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) disease activity score of greater than or equal to (>=) 4 points (with increased deoxyribonucleic acid [DNA] binding item of SLEDAI-2K score based on the ANA Multi-Lyte® ANA-II Plus Test System); 2) no worsening in Physician Global Assessment (MDGA) (worsening is defined as an increase of >=0.3 from baseline on a 0-3 visual analogue scale) and 3) no worsening in British Isles Lupus Assessment Group (BILAG-2004) (worsening is defined as at least 1 new 'A' score or 2 new 'B' scores on the BILAG-2004 compared with baseline).
Time Frame: Day 365
Population: The modified intent-to-treat (mITT) population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 108 | 108 | 108 | 107
percentage of participants | 45.4 | 58.3 | 56.5 | 59.8
Statistical Analysis 1: Comparison: Placebo vs Sifalimumab 200 Milligram (mg); Test type: Superiority or Other; p = 0.057, Regression, Logistic; Odds Ratio (OR) = 1.71, 90% CI 2-sided [1.03 to 2.71]
Statistical Analysis 2: Comparison: Placebo vs Sifalimumab 600 mg; Test type: Superiority or Other; p = 0.094, Regression, Logistic; Odds Ratio (OR) = 1.60, 90% CI 2-sided [1.01 to 2.54]
Statistical Analysis 3: Comparison: Placebo vs Sifalimumab 1,200 mg; Test type: Superiority or Other; p = 0.031, Regression, Logistic; Odds Ratio (OR) = 1.84, 90% CI 2-sided [1.16 to 2.94]

2. Primary Outcome: Percentage of Participants Achieving a Positive Response in SRI (4) in 4-Gene Interferon Test High Participants
Description: SRI (4) responder is defined as: 1) a reduction in baseline SLEDAI-2K disease activity score of >=4 points (with increased DNA binding item of SLEDAI-2K score based on the ANA Multi-Lyte® ANA-II Plus Test System); 2) no worsening in Physician Global Assessment (MDGA) (worsening is defined as an increase of >=0.3 from baseline on a 0-3 visual analogue scale) and 3) no worsening in BILAG-2004 (worsening is defined as at least 1 new 'A' score or 2 new 'B' scores on the BILAG-2004 compared with baseline).
Time Frame: Day 365
Population: The mITT population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement. Here, "N" signifies number of participants with positive diagnostic test.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 88 | 87 | 88 | 87
percentage of participants | 42.0 | 57.5 | 50.0 | 57.5
Statistical Analysis 1: Comparison: Placebo vs Sifalimumab 200 Milligram (mg); Test type: Superiority or Other; p = 0.042, Regression, Logistic; Odds Ratio (OR) = 1.88, 90% CI 2-sided [1.13 to 3.14]
Statistical Analysis 2: Comparison: Placebo vs Sifalimumab 600 mg; Test type: Superiority or Other; p = 0.264, Regression, Logistic; Odds Ratio (OR) = 1.41, 90% CI 2-sided [0.85 to 2.35]
Statistical Analysis 3: Comparison: Placebo vs Sifalimumab 1,200 mg; Test type: Superiority or Other; p = 0.038, Regression, Logistic; Odds Ratio (OR) = 1.91, 90% CI 2-sided [1.14 to 3.19]

3. Secondary Outcome: Percentage of Participants on Greater Than or Equal to 10 mg/Day Oral Prednisone (or Equivalent) at Baseline Who Were Able to Reduce to Less Than or Equal to (<=) 7.5 mg/Day
Description: Percentage of participants on >=10 mg/day oral corticosteroids (OCS) at baseline who were able to taper it to <=7.5 mg/day by Day 365 were recorded.
Time Frame: Day 365
Population: The mITT population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement. Here, "N" signifies number of participants on >=10 mg/day oral prednisone (or equivalent) at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 62 | 61 | 53 | 65
percentage of participants
  Reduce OCS to <=7.5 mg/day: Yes | 6.5 | 8.2 | 9.4 | 6.2
  Reduce OCS to <=7.5 mg/day: No | 93.5 | 91.8 | 90.6 | 93.8
Statistical Analysis 1: Comparison: Placebo vs Sifalimumab 200 Milligram (mg); Test type: Superiority or Other; p = 0.808, Regression, Logistic; Odds Ratio (OR) = 1.19, 90% CI 2-sided [0.37 to 3.81]
Statistical Analysis 2: Comparison: Placebo vs Sifalimumab 600 mg; Test type: Superiority or Other; p = 0.598, Regression, Logistic; Odds Ratio (OR) = 1.45, 90% CI 2-sided [0.45 to 4.66]
Statistical Analysis 3: Comparison: Placebo vs Sifalimumab 1,200 mg; Test type: Superiority or Other; p = 0.884, Regression, Logistic; Odds Ratio (OR) = 0.90, 90% CI 2-sided [0.27 to 3.02]

4. Secondary Outcome: Percentage of Participants With a Cutaneous Lupus Erythematosus Disease Activity and Severity Index (CLASI) Activity Score Greater Than or Equal to (>=) 10 at Baseline Who Achieved a >= 4-point Reduction
Description: The CLASI consists of two scores, the first summarizes the activity of the disease while the second is a measure of the damage done by the disease. Activity is scored on the basis of erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. Damage is scored in terms of dyspigmentation and scarring, including scarring alopecia. The percentage of participants with a CLASI activity score >=10 at baseline who achieved a clinically significant (>=4-point) reduction at Day 365 were reported.
Time Frame: Day 365
Population: The mITT population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement. Here, "N" signifies number of participants with a CLASI activity score >=10 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 35 | 33 | 33 | 26
percentage of participants
  Achieved >=4-point reduction: Yes | 48.6 | 72.7 | 57.6 | 73.1
  Achieved >=4-point reduction: No | 51.4 | 27.3 | 42.4 | 26.9
Statistical Analysis 1: Comparison: Placebo vs Sifalimumab 200 Milligram (mg); Test type: Superiority or Other; p = 0.044, Regression, Logistic; Odds Ratio (OR) = 2.92, 90% CI 2-sided [1.22 to 7.01]
Statistical Analysis 2: Comparison: Placebo vs Sifalimumab 600 mg; Test type: Superiority or Other; p = 0.498, Regression, Logistic; Odds Ratio (OR) = 1.40, 90% CI 2-sided [0.62 to 3.19]
Statistical Analysis 3: Comparison: Placebo vs Sifalimumab 1,200 mg; Test type: Superiority or Other; p = 0.049, Regression, Logistic; Odds Ratio (OR) = 3.03, 90% CI 2-sided [1.20 to 7.68]

5. Secondary Outcome: Percentage of Participants Who Achieved a Greater Than 3-Point Improvement in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Day 365
Population: The mITT population included all randomized participants who received any investigational product and had a baseline primary efficacy measurement. Here, "N" signifies number of participants with a FACIT-fatigue score <49 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 105 | 105 | 102 | 101
percentage of participants
  Achieved > 3-point improvement: Yes | 30.5 | 38.1 | 42.2 | 35.6
  Achieved > 3-point improvement: No | 69.5 | 61.9 | 57.8 | 64.4
Statistical Analysis 1: Comparison: Placebo vs Sifalimumab 200 Milligram (mg); Test type: Superiority or Other; p = 0.270, Regression, Logistic; Odds Ratio (OR) = 1.39, 90% CI 2-sided [0.85 to 2.25]
Statistical Analysis 2: Comparison: Placebo vs Sifalimumab 600 mg; Test type: Superiority or Other; p = 0.077, Regression, Logistic; Odds Ratio (OR) = 1.69, 90% CI 2-sided [1.04 to 2.74]
Statistical Analysis 3: Comparison: Placebo vs Sifalimumab 1,200 mg; Test type: Superiority or Other; p = 0.453, Regression, Logistic; Odds Ratio (OR) = 1.25, 90% CI 2-sided [0.76 to 2.05]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent defined as events present at baseline that worsened in intensity after administration of investigational product or events absent at baseline that emerged after administration of investigational product, for the period extending until the end of participant participation in the study.
Time Frame: Day 1 up to Week 74
Population: The safety population included all participants who received any investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 108 | 108 | 108 | 107
participants
  TEAE | 94 | 97 | 97 | 93
  TESAE | 19 | 16 | 22 | 21

7. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Laboratory investigations included hematology, serum chemistries and urinalysis parameters. Participants with clinically significant abnormalities in these laboratory investigations recorded as TEAEs were reported.
Time Frame: Day 1 up to Week 61
Population: The safety population included all participants who received any investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 108 | 108 | 108 | 107
participants
  Anaemia | 1 | 4 | 4 | 2
  White blood cell count increased | 3 | 1 | 2 | 3
  Neutrophil count increased | 3 | 1 | 2 | 2
  Iron deficiency anaemia | 1 | 2 | 0 | 2
  Haemoglobin decreased | 0 | 1 | 0 | 1
  Lymphocyte count decreased | 2 | 1 | 1 | 0
  White blood cell count decreased | 1 | 0 | 1 | 1
  Autoimmune haemolytic anaemia | 1 | 1 | 0 | 0
  Eosinophilia | 0 | 0 | 0 | 1
  Haematocrit increased | 0 | 0 | 1 | 0
  Haemoglobin increased | 0 | 0 | 1 | 0
  Leukopenia | 0 | 1 | 0 | 0
  Lymphopenia | 1 | 1 | 0 | 0
  Neutropenia | 3 | 0 | 0 | 1
  Neutrophil count decreased | 1 | 0 | 0 | 1
  Platelet count increased | 0 | 0 | 1 | 0
  Red blood cell count decreased | 0 | 0 | 0 | 1
  Thrombocytopenia | 0 | 1 | 0 | 0
  Platelet count decreased | 2 | 0 | 0 | 0
  Monocyte count increased | 1 | 0 | 0 | 0
  Hypokalaemia | 4 | 1 | 4 | 5
  Alanine aminotransferase increased | 5 | 1 | 1 | 3
  Gamma-glutamyltransferase increased | 5 | 0 | 1 | 4
  Hypertriglyceridaemia | 2 | 1 | 1 | 3
  Dyslipidaemia | 2 | 0 | 2 | 2
  Hepatic enzyme increased | 2 | 2 | 2 | 0
  Aspartate aminotransferase increased | 2 | 1 | 0 | 2
  Blood creatine phosphokinase increased | 2 | 0 | 2 | 0
  Blood creatinine increased | 0 | 1 | 0 | 1
  Blood glucose increased | 1 | 0 | 0 | 2
  Hyperglycaemia | 1 | 0 | 0 | 2
  Transaminases increased | 1 | 0 | 1 | 1
  Blood potassium decreased | 0 | 1 | 1 | 0
  Low density lipoprotein increased | 0 | 1 | 1 | 0
  Blood albumin decreased | 0 | 0 | 1 | 0
  Blood alkaline phosphatase decreased | 1 | 0 | 0 | 1
  Blood calcium increased | 1 | 0 | 1 | 0
  Blood cholesterol increased | 0 | 0 | 1 | 0
  Blood homocysteine increased | 0 | 0 | 1 | 0
  Liver function test abnormal | 1 | 0 | 1 | 0
  Hyperlipidaemia | 0 | 0 | 0 | 1
  Hypoalbuminaemia | 2 | 0 | 1 | 0
  Hypoglycaemia | 0 | 0 | 0 | 1
  Blood bilirubin increased | 1 | 0 | 0 | 0
  Hypocalcaemia | 1 | 0 | 0 | 0
  Blood triglycerides increased | 1 | 0 | 1 | 0
  Hyperbilirubinaemia | 0 | 0 | 1 | 0
  Hypertransaminasaemia | 0 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included blood pressure, pulse rate, temperature, weight and respiratory rate. Vital signs abnormalities recorded as TEAEs were reported.
Time Frame: Day 1 up to Week 61
Population: The safety population included all participants who received any investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 108 | 108 | 108 | 107
participants
  Pyrexia | 3 | 2 | 6 | 7
  Hypertension | 7 | 4 | 5 | 4
  Weight increased | 0 | 1 | 2 | 2
  Blood pressure increased | 1 | 2 | 1 | 0
  Chills | 1 | 2 | 0 | 1
  Hypertensive crisis | 0 | 0 | 0 | 1
  Orthostatic hypotension | 1 | 0 | 0 | 1
  Weight decreased | 1 | 0 | 0 | 1
  Hypotension | 1 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings Reported as TEAEs
Description: The 12-lead ECG data were summarized and evaluated. Number of participants with clinically significant abnormal ECG findings as assessed by cardiologist were recorded and reported as TEAEs.
Time Frame: Day 1 up to Week 56
Population: The safety population included all participants who received any investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Sifalimumab 200 Milligram (mg) | Sifalimumab 600 mg | Sifalimumab 1,200 mg
Number analyzed (Participants) | 108 | 108 | 108 | 107
participants | 2 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 74
Description: TEAE defined as events present at baseline that worsened in intensity after administration of investigational product or events absent at baseline that emerged after administration of investigational product, for the period extending until the end of participant participation in the study.
Groups:
- Placebo: Placebo matching to sifalimumab administered intravenously for 48 weeks (Day 337).
- Sifalimumab 200 mg: Sifalimumab 200 milligram (mg) administered intravenously for 48 weeks (Day 337).
- Sifalimumab 600 mg: Sifalimumab 600 mg administered intravenously for 48 weeks (Day 337).
- Sifalimumab 1200 mg: Sifalimumab 1,200 mg administered intravenously for 48 weeks (Day 337).
Arm/Group | Placebo | Sifalimumab 200 mg | Sifalimumab 600 mg | Sifalimumab 1200 mg
Serious Adverse Events (participants affected / at risk) | 19/108 | 16/108 | 22/108 | 21/107
Other Adverse Events (participants affected / at risk) | 93/108 | 94/108 | 96/108 | 92/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | Sifalimumab 200 mg (N=108) | Sifalimumab 600 mg (N=108) | Sifalimumab 1200 mg (N=107)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Corneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ludwig angina (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Septic embolus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 7 (9) | 3 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic limb pain (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | Sifalimumab 200 mg (N=108) | Sifalimumab 600 mg (N=108) | Sifalimumab 1200 mg (N=107)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (7) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 1 (1) | 5 (5) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 7 (7) | 9 (9) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (12) | 4 (5) | 7 (11) | 5 (7)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 6 (8) | 3 (3)
Pyrexia (General disorders) | 3 (4) | 2 (3) | 6 (10) | 7 (10)
Bronchitis (Infections and infestations) | 8 (8) | 11 (15) | 4 (7) | 15 (20)
Conjunctivitis (Infections and infestations) | 4 (5) | 4 (5) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 5 (6) | 5 (6) | 5 (6) | 4 (4)
Herpes zoster (Infections and infestations) | 1 (1) | 5 (6) | 4 (4) | 8 (8)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 10 (17) | 12 (14) | 13 (15) | 9 (12)
Oral herpes (Infections and infestations) | 5 (6) | 3 (7) | 3 (4) | 4 (5)
Pharyngitis (Infections and infestations) | 4 (5) | 3 (3) | 6 (9) | 12 (12)
Respiratory tract infection (Infections and infestations) | 3 (5) | 1 (1) | 3 (3) | 3 (4)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 10 (16) | 17 (27) | 15 (23)
Urinary tract infection (Infections and infestations) | 14 (19) | 22 (25) | 17 (22) | 18 (25)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 3 (3) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (10) | 8 (17) | 7 (9) | 5 (10)
Alanine aminotransferase increased (Investigations) | 5 (7) | 1 (1) | 1 (1) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 5 (7) | 0 (0) | 1 (2) | 4 (5)
White blood cell count increased (Investigations) | 3 (4) | 1 (1) | 2 (4) | 3 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (4) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 4 (5) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (3) | 9 (11) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 8 (8) | 5 (5)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 35 (56) | 34 (42) | 31 (46) | 26 (46)
Dizziness (Nervous system disorders) | 5 (5) | 5 (6) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 15 (24) | 16 (18) | 15 (37) | 12 (13)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (6) | 2 (2) | 7 (8)
Insomnia (Psychiatric disorders) | 4 (4) | 7 (8) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 5 (5) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (8) | 3 (3) | 5 (8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 7 (8) | 4 (4) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.